CLINICAL TRIAL: NCT00560001
Title: Medication Dispenser: MD2: Improving Health Outcomes
Brief Title: MD.2 Medication Dispenser Medication Adherence Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Interactive Medical Developments (Industry)
Collaborators: University of Iowa (Other); Department of Health and Human Services (U.S. Federal Agency); National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PHS 2003-2 FAST TRACK; 5R42AG021844-02 (NIH)
Record Dates: First submitted 2007-11-15; First posted 2007-11-19 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2007-11

CONDITIONS: Frail Elderly; Medication Errors
Keywords: frail elderly; medication errors; patient compliance & attitudes; guideline adherence
MeSH Terms: conditions — Patient Compliance; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Those subjects that receive an MD.2 Medication Dispenser
  Interventions: Behavioral: MD.2 Medication Dispenser
- B (No Intervention): Control subjects that do not receive an MD.2 Medication Dispenser, but continue to take their medications utilizing standard care, such as pill boxes, etc.
  Interventions: Behavioral: MD.2 Medication Dispenser

INTERVENTIONS:
Behavioral: MD.2 Medication Dispenser — For those subjects receiving an MD.2 Medication Dispenser, the machine organizes medications and provides verbal and auditory explicit reminders for individuals to take their medications. At the scheduled time, the patient gets a series of reminders. The patient is then expected to push a single button to dispense a pre-filled medication cup. An automatic record is kept of the subject's medication adherence. Interviewer-administered surveys of the Geriatric Depression Scale, SF-12 Health Status Inventory, self-reported medication compliance and recent hospitalizations and emergency room visits will be given. Caregivers will complete the Caregiver Burden Interview.

SUMMARY:
The objective of this study is to quantify the benefits of using the MD.2 on health outcomes.

DETAILED DESCRIPTION:
A sizeable portion of admissions to hospital and even nursing homes can be avoided if individuals with medication management problems were provided assistive devices to assist with their medications. The MD.2 medication dispenser and monitoring system was developed by Interactive Medical Developments LC and may offer increased support to the elderly with fewer human resources and a substantially reduced cost to the public health system. A rigorous evaluation of this technology has not been conducted. The objective of this Phase III clinical trial (Phase II of this STTR Fast Track Application) is to quantify the benefits of using the MD.2 on health outcomes. The specific aims are to: (1) Quantify healthcare utilization including hospitalizations and emergency room visits for MD.2 clients compared to control clients, (2) Determine the length of time in case management for MD.2 clients compared to control clients, (3) Measure changes in caregiver burden between those with the MD.2 and those with usual medication routines and (4) Determine if cognitive and functional characteristics influence compliance rates among the MD.2 clients and control clients. This study will be conducted in all counties in four of the Area Agencies on Aging in Iowa (who participated in the Phase I study), with the Veteran's Administration(VA)in Iowa, and with Area Agencies on Aging in Illinois. One hundred and fifty clients will be randomized to receive the MD.2 and 150 clients will be randomized to the control group. Primary caregivers for these 300 subjects will also be recruited. Nurses employed by Interactive Medical Developments LC will collect all data. From homecare charts/claims, age, sex, residence, living status, social support, activities of daily living, instrumental activities of daily living, cognition, medical conditions and medication lists will be obtained. Enrolled subjects will also complete an interviewer-administered survey of the Geriatric Depression Scale, SF-12 Health Status Inventory, self-reported medication compliance and recent hospitalizations and emergency room visits. Caregivers will complete the Caregiver Burden Interview. Poisson regression and Cox proportional hazards models will be the primary statistical approaches.

ELIGIBILITY:
Inclusion Criteria:

A client must:

* Be coming up for regular review in Case or Medication Management
* Require medication management services
* Have two or more doses of medication per day
* Have someone to fill MD.2
* Be in independent living (may be assisted living with NO medication management services)
* Be expected to live through follow-up period of six months
* Have an active phone line that can be utilized by the MD.2 system.

Exclusion Criteria:

A client cannot have/or be the following:

* Have someone available to administer medications for every dose
* Have someone in household who is likely to interfere with MD.2
* Blind AND deaf
* Eligible for hospice
* An MD.2 currently

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2006-01; Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
The rate of hospitalizations and emergency room visits will be compared between the MD.2 and control clients | per month (30 client days) over 6 consecutive months

SECONDARY OUTCOMES:
Compare the length of time in case management for MD.2 clients to control clients. | Over 6 consecutive months.
Measure changes in caregiver stressors and burden between those with the MD.2 and those with their usual medication routine. | Over 6 consecutive months
Determine if cognitive and functional characteristics influence compliance rates among the frail elderly using the MD.2. | Over 6 consecutive months

CONTACTS AND LOCATIONS:
Overall Officials: Karen Farris, Ph.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Background] Stuck AE, Beers MH, Steiner A, Aronow HU, Rubenstein LZ, Beck JC. Inappropriate medication use in community-residing older persons. Arch Intern Med. 1994 Oct 10;154(19):2195-200. PMID 7944840
- [Background] Aparasu RR, Mort JR. Inappropriate prescribing for the elderly: beers criteria-based review. Ann Pharmacother. 2000 Mar;34(3):338-46. doi: 10.1345/aph.19006. PMID 10917382
- [Background] Zhan C, Sangl J, Bierman AS, Miller MR, Friedman B, Wickizer SW, Meyer GS. Potentially inappropriate medication use in the community-dwelling elderly: findings from the 1996 Medical Expenditure Panel Survey. JAMA. 2001 Dec 12;286(22):2823-9. doi: 10.1001/jama.286.22.2823. PMID 11735757
- [Background] Gray SL, Mahoney JE, Blough DK. Adverse drug events in elderly patients receiving home health services following hospital discharge. Ann Pharmacother. 1999 Nov;33(11):1147-53. doi: 10.1345/aph.19036. PMID 10573310
- [Background] Kimura H. Effects of caffeine on cleavage delay of sea urchin eggs induced by ethidium bromide or puromycin. J Radiat Res. 1975 Jun;16(2):125-31. doi: 10.1269/jrr.16.125. No abstract available. PMID 1171974
- [Background] Bero LA, Lipton HL, Bird JA. Characterization of geriatric drug-related hospital readmissions. Med Care. 1991 Oct;29(10):989-1003. doi: 10.1097/00005650-199110000-00005. PMID 1921531
- [Background] Chrischilles EA, Segar ET, Wallace RB. Self-reported adverse drug reactions and related resource use. A study of community-dwelling persons 65 years of age and older. Ann Intern Med. 1992 Oct 15;117(8):634-40. doi: 10.7326/0003-4819-117-8-634. PMID 1530194
- [Background] Farris KD, Kelly MW, Tryon J. Clock drawing test and medication complexity index as indicators of medication management capacity: a pilot study. J Am Pharm Assoc (Wash). 2003 Jan-Feb;43(1):78-81. No abstract available. PMID 12585756
- [Background] Col N, Fanale JE, Kronholm P. The role of medication noncompliance and adverse drug reactions in hospitalizations of the elderly. Arch Intern Med. 1990 Apr;150(4):841-5. PMID 2327844
- [Background] DiMatteo MR, Giordani PJ, Lepper HS, Croghan TW. Patient adherence and medical treatment outcomes: a meta-analysis. Med Care. 2002 Sep;40(9):794-811. doi: 10.1097/00005650-200209000-00009. PMID 12218770
- [Background] Buckwalter KC, Wakefield BJ, Hanna B, Lehmann J. New technology for medication adherence: electronically managed medication dispensing system. J Gerontol Nurs. 2004 Jul;30(7):5-8. doi: 10.3928/0098-9134-20040701-04. No abstract available. PMID 15287321
- [Background] Maddigan SL, Farris KB, Keating N, Wiens CA, Johnson JA. Predictors of older adults' capacity for medication management in a self-medication program: a retrospective chart review. J Aging Health. 2003 May;15(2):332-52. doi: 10.1177/0898264303251893. PMID 12795276
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086